CLINICAL TRIAL: NCT01097707
Title: A Phase 2 Clinical Study to Evaluate Daily Oral Doses of LY500307 for 24 Weeks in Men With Lower Urinary Tract Symptoms (LUTS) and Prostatic Enlargement Secondary to Benign Prostatic Hyperplasia (BPH)
Brief Title: A Study in Men With Benign Prostatic Hyperplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10373; I1A-MC-BPAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — erteberel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1mg LY500307 (Experimental)
  Interventions: Drug: LY500307
- 3mg LY500307 (Experimental)
  Interventions: Drug: LY500307
- 10mg LY500307 (Experimental)
  Interventions: Drug: LY500307
- 25mg LY500307 (Experimental)
  Interventions: Drug: LY500307
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY500307 — Administered orally, daily for 24 weeks
  Arms: 10mg LY500307; 1mg LY500307; 25mg LY500307; 3mg LY500307
Drug: Placebo — Administered orally, daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether LY500307 helps symptoms of Benign Prostatic Hyperplasia (BPH)

ELIGIBILITY:
Inclusion Criteria:

* Present at screening with a history of benign prostatic hyperplasia (BPH) for >6 months.
* Have an International Prostate Symptom Score (IPSS) greater than or equal to 13 at screening.
* Have a total prostate volume by transrectal ultrasound greater than or equal to 30 milliliter (mL) at screening.
* Show signs of bladder outlet obstruction as defined by a peak urinary flow rate (Qmax) greater than or equal to 4 and less than or equal to 15 milliliter/second (mL/sec) (from a prevoid total bladder volume [assessed by ultrasound] of greater than or equal to 150 to less than or equal to 550 ml and a minimum voided volume of 125 ml) at screening.
* Have a prostate-specific antigen (PSA) greater than or equal to 1.4 and less than or equal to 10 nanogram/milliliter (ng/mL) at screening.
* Demonstrate a Post Void Residual less than or equal to 300 mL by ultrasound at screening.
* Have not received the following treatments within the specified time period:

  1. Finasteride or dutasteride for at least 6 months prior to screening.
  2. Any alpha-adrenergic antagonists for at least 4 weeks prior to screening.
  3. Any other non-experimental BPH therapy (including an herbal preparation) for at least 4 weeks prior to screening.
  4. Any other experimental or off-label BPH therapy such as injectable therapies with a protracted effect for at least 6 months prior to screening.
  5. Any overactive bladder treatment for at least 4 weeks prior to screening.
  6. Any Erectile Dysfunction treatment which may include oral phosphodiesterase type 5 inhibitors or devices for at least 4 weeks prior to screening.
* Have a morning fasting Total Testosterone concentration greater than or equal to 300 nanogram/deciliter (ng/dL) at screening.
* If hyperlipidemic, based on history, be stable on statin treatment as determined by the investigator for at least 2 months prior to screening.

Exclusion Criteria:

* Have completed or withdrawn from this study or have completed or withdrawn from any other study investigating LY500307.
* Have any history of BPH-related invasive procedures (for example, Transurethral Resection of the Prostate, open prostatectomy, and minimally invasive procedures that include thermal-based therapies, transurethral microwave treatment, transurethral needle ablation, and stents).
* Have active cardiovascular disease as evidenced by the following:

  1. Recent Myocardial infarction, unstable angina, stroke or Transient ischemic attack within 6 months of screening.
  2. Recent coronary intervention that includes coronary artery bypass surgery, percutaneous coronary artery intervention, or stent placement within 6 months of screening.
  3. Recent history of positive stress tests without any written documentation of effective intervention within 6 months of screening.
  4. Evidence of heart disease categorized as greater than or equal to Class III functional classification of New York Heart Association (NYHA) within 6 months of screening.
* Have known or suspected history of prostate cancer, breast cancer, or other clinically significant neoplastic disease (other than squamous cell or basal cell carcinoma of skin).
* Have a history of deep venous thrombosis or pulmonary embolism disease.
* Have moderate to severe renal insufficiency.
* Have a hemoglobin A1c (HbA1c) greater than 9.0%.
* Are on testosterone replacement therapy, or drugs that influence the hypothalamus-pituitary-gonadal axis.
* Are on pharmacological treatment other than statins for hyperlipidemia.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (40):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendora, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Bernardino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarzana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parker, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlebury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Celebration, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coeur d'Alene, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbelt, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poughkeepsie, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmond, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bala-Cynwyd, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bentleigh East, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mentone, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint John, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garches
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Bergzaben
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holzminden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oranienburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reutlingen
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cefalà Diana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg LY500307; 3 mg LY500307; 10 mg LY500307; 25 mg LY500307: LY500307: Administered orally, daily for 24 weeks
Period: Overall Study
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Started | 83 | 80 | 82 | 84 | 85
Completed | 39 | 37 | 37 | 40 | 35
Not Completed | 44 | 43 | 45 | 44 | 50
Not completed — Abnormal Lab/Electrocardiogram Result | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 4 | 2 | 3 | 1 | 3
Not completed — Entry Criteria Not Met | 2 | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 3
Not completed — Protocol Violation | 2 | 2 | 3 | 2 | 2
Not completed — Sponsor Decision | 31 | 31 | 34 | 35 | 36
Not completed — Withdrawal by Subject | 3 | 6 | 1 | 4 | 3
Not completed — Reason unknown | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo | Total
Number analyzed (Participants) | 83 | 80 | 82 | 84 | 85 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.97 (7.55) | 67.67 (7.34) | 67.21 (7.10) | 63.18 (7.34) | 64.11 (7.92) | 65.80 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 83 | 80 | 82 | 84 | 85 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 4 | 1 | 12
  Not Hispanic or Latino | 79 | 79 | 80 | 80 | 84 | 402
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 2 | 0 | 5 | 14
  White | 78 | 75 | 79 | 82 | 80 | 394
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 2 | 2 | 2 | 2 | 3 | 11
  United States | 42 | 41 | 41 | 43 | 42 | 209
  Canada | 5 | 5 | 5 | 5 | 6 | 26
  Greece | 2 | 1 | 2 | 2 | 2 | 9
  Australia | 3 | 3 | 3 | 3 | 3 | 15
  Russia | 12 | 12 | 12 | 12 | 13 | 61
  Germany | 12 | 11 | 12 | 12 | 11 | 58
  Italy | 5 | 5 | 5 | 5 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24-Week Endpoint in International Prostate Symptom Score (IPSS) Total Score
Description: IPSS Total Score is the sum of Questions 1 through 7 of the IPSS questionnaire. Each question is scored from 0 (none/no symptoms) to 5 (frequent symptoms) with an IPSS Total Score range of 0-35 points. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline IPSS total score measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 44 | 44 | 47 | 50 | 45
units on a scale | -1.34 (6.56) | -2.61 (7.00) | -3.68 (6.69) | -4.38 (5.68) | -3.44 (6.82)

2. Secondary Outcome: Percentage Change From Baseline to 24-Week Endpoint in Total Prostate Volume (TPV)
Description: The TPV measurement (milliliters) by transrectal ultrasound (TRUS) is an established diagnostic test for men with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH).
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline TPV measurement.
Measure: Mean (Standard Deviation); unit: percentage change in TPV
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 44 | 44 | 46 | 49 | 44
percentage change in TPV | 1.6 (22.7) | -4.5 (15.6) | -6.7 (17.2) | 1.3 (20.6) | -6.6 (15.5)

3. Secondary Outcome: Change From Baseline to 24-Week Endpoint in Peak Urinary Flow Rate (Qmax)
Description: Qmax is defined as the peak urine flow rate measured using standard calibrated uroflowmeter.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline Qmax measurement.
Measure: Mean (Standard Deviation); unit: milliliters/second (mL/sec)
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 40 | 36 | 41 | 38 | 37
milliliters/second (mL/sec) | 0.76 (3.60) | 1.53 (4.47) | 0.87 (2.95) | 0.11 (3.51) | 1.32 (5.42)

4. Secondary Outcome: Change From Baseline to 24-Week Endpoint in International Prostate Symptom Score-Quality of Life Index (IPSS-QoL)
Description: IPSS QoL assesses participant's response to the following question: "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response options are Delighted (0), Pleased (1); Mostly satisfied (2); Mixed-about equally satisfied and dissatisfied (3); Mostly dissatisfied (4); Unhappy (5); Terrible (6), with a total range of 0-6.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline IPSS-QoL measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 44 | 44 | 48 | 50 | 45
units on a scale | -0.27 (1.25) | -0.75 (1.28) | -0.60 (1.18) | -0.82 (1.21) | -0.71 (1.08)

5. Secondary Outcome: Change From Baseline to 24-Week Endpoint in International Prostate Symptom Score (IPSS) Storage, Voiding and Nocturia Subscores
Description: IPSS Storage (Irritative) subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores range from 0 (no irritative symptoms) to 5 (frequent irritative symptoms), with a total subscore of the 3 questions for irritative subscore ranging from 0 to 15. IPSS Voiding (Obstructive) subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 0 (no obstructive symptoms) to 5 (frequent obstructive symptoms), with a total subscore of the 4 questions of the obstructive score ranging from 0 to 20. Nocturia Subscore is IPSS Question 7, which assesses how many times over the last month a participant gets up to urinate from the time they went to bed at night until the time they got up in the morning. Scores range from 0=None; 1=1 time; 2= 2 times; 3=3 times; 4=4 times; 5=5 or more times.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline IPSS subscores measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 44 | 44 | 48 | 50 | 45
units on a scale
  IPSS storage subscore: number analyzed (Participants) | 44 | 44 | 47 | 50 | 45
  IPSS storage subscore | -0.73 (3.49) | -0.82 (3.66) | -1.64 (3.19) | -1.86 (2.92) | -1.47 (3.35)
  IPSS voiding subscore: number analyzed (Participants) | 44 | 44 | 47 | 50 | 45
  IPSS voiding subscore | -0.61 (3.69) | -1.80 (4.81) | -2.04 (4.09) | -2.52 (3.72) | -1.98 (4.34)
  IPSS Nocturia subscore | -0.23 (1.34) | -0.16 (1.49) | -0.54 (1.20) | -0.54 (1.58) | -0.47 (1.29)

6. Secondary Outcome: Percentage Change From Baseline to 24-Week Endpoint in Prostate Specific Antigen (PSA)
Description: The units of PSA measurement are nanograms per milliliter (ng/mL).
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline PSA measurement.
Measure: Mean (Standard Deviation); unit: percentage change in PSA
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 55 | 59 | 59 | 65 | 56
percentage change in PSA | 18.81 (47.00) | 6.62 (31.55) | 14.34 (36.30) | 5.66 (27.32) | 8.65 (50.67)

7. Secondary Outcome: Change From Baseline to 24-Week Endpoint in Fasting Total Testosterone
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline fasting total testosterone measurement.
Measure: Mean (Standard Deviation); unit: nanogram/deciliter (ng/dL)
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 54 | 57 | 59 | 63 | 57
nanogram/deciliter (ng/dL) | -12.5 (166.4) | -1.3 (129.6) | -24.9 (112.2) | 24.6 (136.7) | -14.6 (122.7)

8. Secondary Outcome: Change From Baseline to 24-Week Endpoint in Lipid Profile
Description: The lipid profile consisted of low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides.
Time Frame: Baseline, 24 weeks
Population: All randomized participants who had baseline and one post-baseline lipid measurement.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Number analyzed (Participants) | 55 | 59 | 60 | 65 | 58
milligram/deciliter (mg/dL)
  LDL-C: number analyzed (Participants) | 54 | 56 | 59 | 64 | 57
  LDL-C | -0.4 (22.5) | -1.8 (20.3) | -1.1 (27.3) | -12.6 (87.7) | 3.6 (21.9)
  HDL-C: number analyzed (Participants) | 55 | 58 | 60 | 65 | 58
  HDL-C | -0.98 (5.93) | 1.11 (6.83) | 0.42 (9.31) | 1.23 (7.13) | 0.16 (7.63)
  Triglyceride | 3.91 (103.66) | -0.71 (45.84) | 6.61 (62.33) | -2.15 (66.69) | 2.23 (62.99)

ADVERSE EVENTS:
Arm/Group | 1 mg LY500307 | 3 mg LY500307 | 10 mg LY500307 | 25 mg LY500307 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/83 | 3/80 | 3/82 | 2/84 | 3/85
Other Adverse Events (participants affected / at risk) | 32/83 | 32/80 | 31/82 | 30/84 | 37/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg LY500307 (N=83) | 3 mg LY500307 (N=80) | 10 mg LY500307 (N=82) | 25 mg LY500307 (N=84) | Placebo (N=85)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Residual urine volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg LY500307 (N=83) | 3 mg LY500307 (N=80) | 10 mg LY500307 (N=82) | 25 mg LY500307 (N=84) | Placebo (N=85)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Therapeutic response unexpected (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 5 (6) | 6 (6)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood luteinising hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood testosterone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Protein urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Semen analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cells urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymal tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retrograde ejaculation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days